CLINICAL TRIAL: NCT03430349
Title: A Phase 1, Blinded, Single Center Study to Evaluate the Safety and Immunogenicity of Two Novel Live Attenuated Serotype 2 Oral Poliovirus Vaccines, Derived From a Modified Sabin 2 Infectious cDNA Clone, in Healthy Adults Previously Primed With Inactivated Polio Vaccine (IPV)
Brief Title: Phase 1 Novel Live Attenuated Serotype 2 Oral Polio Vaccine Study in Inactivated Polio Vaccine (IPV) Primed Adults
Acronym: nOPV2M4a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Van Damme (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); PATH (Other); Celerion (Industry)
Responsible Party: Sponsor-Investigator, Pierre Van Damme, Full Professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: UAM4a; 2017-000908-21 (EudraCT Number)
Record Dates: First submitted 2018-01-21; First posted 2018-02-12 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Poliomyelitis
Keywords: IPV-primed; adults; vaccination; containment; shedding; genetic stability; safety; neurovirulence; novel polio vaccine candidates
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: the study will be conducted with each candidate vaccine sequentially. After randomization of the first participant of Group 1 the next 14 participants will all be enrolled in the same Group and receive the same nOPV2 candidate and the next 15 participants will be enrolled in the other Group and receive the corresponding nOPV2 candidate. Prior to the start of the study the clinical research organization (CRO) will provide the site with 2 randomization envelopes for the first subject. By randomly choosing 1 of the envelopes first subject will be dedicated to a certain nOPV2 candidate and this will determine the allocation of the next 14 subjects to the same Group.
  Study staff will be blinded in the same way and will be blinded for individual shedding results of the participants of a Group until end of containment of this Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel OPV2 Candidate 1 (Experimental): Participants received one vaccination with novel OPV2 candidate 1 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ 50% cell culture infectious dose units [CCID50]).
  Interventions: Biological: Novel OPV2 candidate 1
- Novel OPV2 Candidate 2 (Experimental): Participants received one vaccination with novel OPV2 candidate 2 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 2

INTERVENTIONS:
Biological: Novel OPV2 candidate 1 — Live-attenuated serotype-2 poliovirus derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells; candidate 1 (S2/cre5/S15domV/rec1/hifi3).
  Modifications included the following:
  * Changes to the viral nucleotide sequence in part of the 5'-untranslated region to improve the genetic stability of this major attenuating determinant of Sabin type-2 to avoid reversion by single nucleotide changes.
  * Two modifications in the polymerase 3D to further improve stability of the attenuation and reduce frequency of recombination events
  * Relocation of a key replication element from the 2C coding region to the 5'-untranslated region, to inhibit recombination.
  Arms: Novel OPV2 Candidate 1
Biological: Novel OPV2 candidate 2 — Live-attenuated serotype-2 poliovirus derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells; candidate 2 (S2/S15domV/CpG40).
  Modifications included the following:
  * Changes to the viral nucleotide sequence in part of the 5'-untranslated region to improve the genetic stability of this major attenuating determinant of Sabin type-2 to avoid reversion by single nucleotide changes.
  * silent non-coding modifications engineered within the capsid (VP1-4) designed to reduce replicative fitness and, potentially, to improve stability of the attenuated phenotype while also reducing transmission.
  Arms: Novel OPV2 Candidate 2

SUMMARY:
This first-in-human (FIH) phase 1 study is designed to evaluate in contained conditions the safety, immunogenicity, shedding, and genetic stability of two novel oral polio vaccine type 2 (nOPV2) vaccine candidates in IPV-primed adults before testing in a larger adult and adolescent (> 15 y of age) population, and then in young children and infants.

DETAILED DESCRIPTION:
Two nOPV2 vaccine candidates have been developed as attenuated serotype 2 polioviruses derived from a modified Sabin 2 infectious complementary deoxyribonucleic acid (cDNA) clone. nOPV2 Candidate 1 (S2/cre5/S15domV/rec1/hifi3) and nOPV2 Candidate 2 (S2/S15domV/CpG40) were generated by modifying the Sabin-2 ribonucleic acid (RNA) sequence to improve phenotypic stability and make the strains less prone to reversion to virulence.

Due to the withdrawal of Sabin monovalent oral polio vaccine type 2 (mOPV2) and prohibition of its use from April 2016 onwards, well before the availability of nOPV2 for clinical testing, Phase 4 trials have been conducted with Sabin mOPV2 to provide control data on safety, immunogenicity, against which data for nOPV2 in subsequent Phase I and II studies will be evaluated and compared. The Phase 4 trials of Sabin mOPV2 were designed to parallel the expected design of the Phase 1 and 2 nOPV2 studies with respect to overall design, inclusion of similar study cohorts. As for these reasons head to head comparison of nOPV2 and mOPV2 is not possible, the overall clinical development plan with the Phase I and II studies was designed taking into consideration the unique situation of OPV2 cessation in April 2016, and the global public health need of a vaccine with lower risk of vaccine-associated paralytic poliomyelitis (VAPP) and vaccine-derived type-2 poliovirus (cVDPV2) (VDPV2) for outbreak response in the post-cessation era.

This first-in-human phase 1 study is designed to evaluate in contained conditions the safety, immunogenicity, shedding and genetic stability of both nOPV2 vaccine candidates in IPV-primed adults before testing in a larger adult and adolescent (> 15 y of age) population, and then in young children and infants.

This Phase 1 study will include 30 IPV-only vaccinated adults to be vaccinated with the study vaccines (15 subjects per candidate vaccine) and followed in contained conditions (28 days) to obtain safety, immunogenicity, shedding and genetic stability data relevant to the decision to advance to future studies with testing in un-contained conditions.

Participants were isolated in a purpose-built containment facility named Poliopolis at the University of Antwerp Hospital (Antwerp, Belgium), to minimize the risk of environmental release of the novel OPV2 candidates. Volunteers were enrolled sequentially in two groups, with each group receiving one of the two vaccine candidates, to avoid cross-contamination, after which they were confined to Poliopolis for 28 days, with further monitoring until end of shedding. A final safety follow-up call (for those no longer shedding) or visit (for those still shedding) was made 42 days after vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, between 18 and 50 years old, extremes included, having received at least 3 doses of IPV in the past (more than 12 months before the start of the study);
2. In good physical and mental health as determined on the basis of medical history, laboratory screening tests and general physical and psychological examination;
3. Female subjects of childbearing potential must agree to the use of an effective method of birth control throughout the study and up to 3 months after vaccine administration;
4. Willing to adhere to the prohibitions and restrictions specified in this protocol;
5. Willing to adhere to the restrictions of containment for duration as specified in the protocol;
6. Informed Consent Form (ICF) signed voluntarily by the subject before any study-related procedure is performed, indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study.

   Furthermore, willing to adhere to following restrictions as long as shedding will be observed at the end of the containment period:
7. No intention to travel to the Netherlands and to polio endemic countries (updated list will be made available at the start of the study);
8. No professional handling of food, catering or food production activities;
9. Not having household or professional contact with known immunosuppressed people or people without full polio vaccination (i.e. complete primary infant immunization series), e.g. babysitting;
10. No neonatal nursing activities or other professional contact with children under 6 months old;

Exclusion Criteria:

1. A condition that, in the opinion of the Investigator, could compromise the well being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements;
2. Ever having received any OPV in the past;
3. Having Crohn's disease or ulcerative colitis or having had major surgery of the gastrointestinal tract involving significant loss or resection of the bowel;
4. A known allergy, hypersensitivity, or intolerance to the study vaccine, or to any of its components or to any antibiotics;
5. Any confirmed or suspected immunosuppressive or immunodeficiency condition (including human immunodeficiency virus [HIV] infection, hepatitis B and C infections or negative for total serum IgA);
6. Chronic administration (i.e., longer than 14 days) of immunosuppressant drugs or other immune-modifying drugs within 6 months prior to the administration of study vaccine or planned use during the study. For instance, for corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg/day (inhaled and topical steroids are allowed whereas intra-articular and epidural injection/administration of steroids are not allowed);
7. Presence of contraindications to administration of the study vaccine on Day 0: acute severe febrile illness deemed by the Investigator to be a contraindication for vaccination or persistent diarrhea or vomiting;
8. Indications of drug abuse or excessive use of alcohol at Day 0;
9. Being pregnant or breastfeeding. Women of childbearing potential will undergo a pregnancy test at Screening (serum) and at Day 0 (urine). Subjects with a positive pregnancy test will be excluded;
10. Participation in another clinical study within 28 days prior to entry in this study or receipt of any investigational product (drug or vaccine) other than the study vaccine within 28 days prior to the administration of study vaccine, or planned use during the study period;
11. Administration of any vaccine other than the study vaccine within 28 days prior to the administration of study vaccine and during the entire study period;
12. Administration of polio vaccine within 12 months before the start of the study;
13. Having had a transfusion of any blood product or application of immunoglobulins within the 4 weeks prior to the administration of study vaccine or during the study;
14. Subject is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, or is a family member of an employee or the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: pierre van damme, MD,PHD, Principal Investigator — centre for the evaluation of vaccination
Locations (1):
- university of Antwerp - centre for the evaluation of vaccination, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
there is no such plan for the moment

REFERENCES:
- [Derived] Van Damme P, De Coster I, Bandyopadhyay AS, Revets H, Withanage K, De Smedt P, Suykens L, Oberste MS, Weldon WC, Costa-Clemens SA, Clemens R, Modlin J, Weiner AJ, Macadam AJ, Andino R, Kew OM, Konopka-Anstadt JL, Burns CC, Konz J, Wahid R, Gast C. The safety and immunogenicity of two novel live attenuated monovalent (serotype 2) oral poliovirus vaccines in healthy adults: a double-blind, single-centre phase 1 study. Lancet. 2019 Jul 13;394(10193):148-158. doi: 10.1016/S0140-6736(19)31279-6. Epub 2019 Jun 4. PMID 31174831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited via local advertising and confined in a purpose-built containment facility at the University of Antwerp Hospital (Antwerp, Belgium) to minimize the risk of environmental release of the vaccine virus. Volunteers included healthy adults previously vaccinated with inactivated polio vaccine (IPV).
Pre-assignment Details: Participants were enrolled sequentially into one of two groups, and received a single dose of one of two novel oral polio vaccine type 2 (nOPV2) candidates. Participants were monitored for adverse events, immune responses, and fecal shedding of the vaccine virus for 28 days. If if shedding continued beyond 28 days participants were asked to further collect stool samples daily on an ambulatory basis until end of shedding.
Period: Overall Study
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Started | 15 | 15
Received nOPV Vaccination | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received a dose of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (7.72) | 33.5 (10.93) | 32.3 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 14 | 28
  Asian | 0 | 0 | 0
  Black | 0 | 1 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events and Severe Adverse Events Throughout the Study
Description: Serious adverse events are medical events that resulted in death, were life-threatening, required admission to hospital, or resulted in notable incapacity of the individual. Adverse events were also graded from mild to severe; Severe adverse events are medical events that prevent normal everyday activities or fever > 39°C; this category does not include serious adverse events.
  Serious adverse events and severe adverse events include both solicited and unsolicited events. Solicited events comprised signs and symptoms that were reported by the participant using a predefined checklist in a diary card, or a fever, as determined by the participant's measurement of their body temperature, for up to 7 days after vaccination. Unsolicited events comprised other signs and symptoms recorded through the end of the study.
  Adverse events were assessed by the investigator for causality as unrelated, unlikely, possibly, or probably related to the vaccination.
Time Frame: From Day 0 up to 42 days
Population: All randomized participants who received a dose of study vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Novel OPV2 Candidate 1: Participants received one vaccination with novel OPV2 candidate 1 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
Participants
  ≥1 serious adverse event | 0 | 0
  ≥1 severe adverse event (AE) | 6 | 9
  ≥1 severe AE probably related to vaccine | 0 | 0
  ≥1 severe AE possibly related to vaccine | 6 | 9
  ≥1 severe AE unlikely related to vaccine | 0 | 0
  ≥1 severe AE unrelated | 0 | 0

2. Primary Outcome: Percentage of Participants With Viral Shedding
Description: Participants provided stool samples for assessment of viral shedding, defined as the presence of type 2-specific poliovirus ribonucleic acid (RNA) in stools. Samples were analyzed by the US Centers for Disease Control and Prevention (CDC; Atlanta, GA, USA) for the presence of type-2 poliovirus genome using a Sabin multiplex real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay of total nucleic acid extracted from stool suspensions (50% weight to volume in cell culture medium).
Time Frame: Days 0, 1, 2, 3, 4, 5, 6, 7, 14, 21, and 28
Population: All randomized participants who received study vaccine with available stool samples at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
percentage of participants
  Day 0: number analyzed (Participants) | 11 | 9
  Day 0 | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 29.9]
  Day 1: number analyzed (Participants) | 13 | 14
  Day 1 | 38.5 [17.7 to 64.5] | 7.1 [1.3 to 31.5]
  Day 2: number analyzed (Participants) | 14 | 13
  Day 2 | 50.0 [26.8 to 73.2] | 53.8 [29.1 to 76.8]
  Day 3: number analyzed (Participants) | 15 | 14
  Day 3 | 100 [79.6 to 100] | 71.4 [45.4 to 88.3]
  Day 4: number analyzed (Participants) | 14 | 14
  Day 4 | 92.9 [68.5 to 98.7] | 42.9 [21.4 to 67.4]
  Day 5: number analyzed (Participants) | 14 | 12
  Day 5 | 92.9 [68.5 to 98.7] | 83.3 [55.2 to 95.3]
  Day 6: number analyzed (Participants) | 14 | 14
  Day 6 | 100 [78.5 to 100] | 64.3 [38.8 to 83.7]
  Day 7: number analyzed (Participants) | 14 | 11
  Day 7 | 100 [78.5 to 100] | 72.7 [43.4 to 90.3]
  Day 14: number analyzed (Participants) | 13 | 13
  Day 14 | 76.9 [49.7 to 91.8] | 23.1 [8.2 to 50.3]
  Day 21: number analyzed (Participants) | 14 | 13
  Day 21 | 64.3 [38.8 to 83.7] | 23.1 [8.2 to 50.3]
  Day 28: number analyzed (Participants) | 11 | 8
  Day 28 | 45.5 [21.3 to 72.0] | 37.5 [13.7 to 69.4]

3. Primary Outcome: Cell Culture Infective Dose of Shed Virus in Virus-positive Stool Samples
Description: In stool samples that were positive for type-2 poliovirus detected by RT-PCR, infectious virus was measured as 50% cell culture infective dose (CCID₅₀) per gram of stool by use of a modification of the World Health Organization (WHO) cell sensitivity assay.
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 14, 21, and 28
Population: All randomized participants who received study vaccine and with type 2 poliovirus-positive stool samples at each time point.
Measure: Median (95% Confidence Interval); unit: log₁₀ (CCID₅₀/g)
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
log₁₀ (CCID₅₀/g)
  Day 1: number analyzed (Participants) | 5 | 1
  Day 1 | 3.22 [2.88 to 4.09] | 4.41 [4.41 to 4.41]
  Day 2: number analyzed (Participants) | 7 | 7
  Day 2 | 3.66 [3.53 to 3.81] | 3.44 [3.00 to 4.03]
  Day 3: number analyzed (Participants) | 15 | 10
  Day 3 | 4.50 [3.69 to 4.69] | 3.52 [3.00 to 4.02]
  Day 4: number analyzed (Participants) | 13 | 6
  Day 4 | 4.16 [3.91 to 4.41] | 3.27 [2.94 to 4.21]
  Day 5: number analyzed (Participants) | 13 | 10
  Day 5 | 3.84 [3.41 to 4.38] | 3.08 [2.91 to 3.20]
  Day 6: number analyzed (Participants) | 14 | 9
  Day 6 | 3.91 [3.71 to 4.24] | 3.53 [2.88 to 3.78]
  Day 7: number analyzed (Participants) | 14 | 8
  Day 7 | 4.05 [3.84 to 4.53] | 3.44 [2.91 to 3.81]
  Day 14: number analyzed (Participants) | 10 | 3
  Day 14 | 3.06 [2.88 to 3.63] | 2.88 [2.78 to 3.97]
  Day 21: number analyzed (Participants) | 9 | 3
  Day 21 | 3.00 [2.84 to 3.38] | 3.19 [3.06 to 3.94]
  Day 28: number analyzed (Participants) | 5 | 3
  Day 28 | 2.91 [2.75 to 3.69] | 3.19 [3.03 to 4.09]

4. Primary Outcome: Time to Shedding Cessation
Description: The time to cessation of shedding was defined as the time interval between administration of vaccine and the date of the first sample negative for type 2 poliovirus shedding (assessed by RT-PCR) after which the following two consecutive samples were also negative.
  Time to cessation of viral shedding was assessed using Kaplan-Meier methods; participants were right-censored if they had not met this endpoint with the last stool sample collected.
Time Frame: Stool samples were collected from the day of vaccination to Day 28 or until shedding cessation; up to 89 days (novel OPV2 candidate 1) and 48 days (novel OPV candidate 2).
Population: All randomized participants who received a dose of study vaccine with at least one type 2 poliovirus-positive stool sample.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
days | 23 [15 to 36] | 12 [1 to 23]

5. Primary Outcome: Shedding Index
Description: A combined index of the prevalence, duration, and quantity of viral shedding in all participants.
  The viral shedding index was calculated for each participant as the mean of log₁₀(CCID₅₀/g) of samples collected 7, 14, 21, and 28 days after vaccine administration, with the lower limit of quantitation (2.75 log₁₀) as an observed value, and all titers in stool samples with negative shedding results (real-time RT-PCR-negative values) contributing 0 to the mean.
Time Frame: Days 7, 14, 21, and 28
Population: All randomized participants who received a dose of study vaccine. Missing values (from missing samples on specific study days) were replaced with values from the days before or after or the average of these two values, as necessary.
Measure: Median (95% Confidence Interval); unit: log₁₀(CCID₅₀/g)
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
log₁₀(CCID₅₀/g) | 2.84 [1.77 to 3.46] | 0.95 [0.70 to 1.57]

6. Secondary Outcome: Number of Participants With Solicited Adverse Events
Description: Adverse events were solicited from the participants by the medical team during the 7 days after vaccination. Solicited events comprised signs and symptoms that were reported with a predefined checklist in a diary card, including headache, fatigue, myalgia, arthralgia, paresthesia, anesthesia, paralysis, nausea, vomiting, diarrhea and abdominal pain, or fever defined as a temperature of 37.5°C or higher.
  Adverse events were graded as mild (easily tolerated), moderate (sufficiently discomforting to interfere with normal everyday activities), or severe (preventing normal everyday activities, or temperatures higher than 39.0°C).
  Adverse events were assessed by the investigator for causality as unrelated, unlikely, possibly, or probably related to the vaccination.
Time Frame: Day 0 to Day 7
Population: All randomized participants who received a dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
Participants
  Any solicited adverse event | 13 | 9
  Mild | 8 | 8
  Moderate | 5 | 1
  Severe | 0 | 0
  Unrelated/Unlikely related to vaccination | 11 | 2
  Probably/Possibly related to vaccination | 4 | 7

7. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited events comprised other signs and symptoms that participants reported through the end of the study. Each unsolicited AE was rated on a 3-point scale of increasing intensity:
  * Grade 1: Mild; an AE that was easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
  * Grade 2: Moderate; an AE that was sufficiently discomforting to interfere with normal everyday activities.
  * Grade 3: Severe; an AE that prevented normal everyday activities.
  Each adverse event was assessed by the investigator for causality as unrelated, unlikely, possibly, or probably related to the vaccination.
Time Frame: From Day 0 up to 42 days
Population: All randomized participants who received a dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
Participants
  Any unsolicited adverse event | 15 | 15
  Mild | 3 | 3
  Moderate | 6 | 3
  Severe | 6 | 9
  Unrelated/Unlikely related to vaccination | 14 | 9
  Probably/Possibly related to vaccination | 10 | 12

8. Secondary Outcome: Number of Participants With Clinically Relevant Deviations From Normal Laboratory Evaluations
Description: Clinical laboratory test values were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (toxicity grades) or in accordance with the normal ranges of the clinical laboratory (below, within, or above normal range) for parameters for which no toxicity grades were defined.
  Clinical chemistry assessments included total bilirubin, glucose, blood urea nitrogen (BUN), creatinine, calcium, inorganic phosphate, potassium, sodium, alanine aminotransferase, aspartate aminotransferase, and C-reactive protein (CRP). Hematology assessments included hemoglobin, hematocrit, red blood cells, and white blood cells with differential.
Time Frame: Screening, Day 7, Day 14, and Day 28
Population: All randomized participants who received study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
Participants
  Clinical Chemistry at Screening | 1 | 0
  Clinical Chemistry at Day 7 | 4 | 7
  Clinical Chemistry at Day 14 | 3 | 5
  Clinical Chemistry at Day 28 | 6 | 1
  Hematology at Screening | 1 | 0
  Hematology at Day 7 | 0 | 1
  Hematology at Day 14 | 0 | 1
  Hematology at Day 28 | 0 | 0

9. Secondary Outcome: Anti-Poliovirus Type-2 Neutralizing Antibody Titers
Description: Neutralizing antibodies against poliovirus type 2 were determined using the WHO standard microneutralization assay (WHO EPI GEN 93.9).
Time Frame: Day 0 and Day 28
Population: All randomized participants who received study vaccine and had no exclusion criterion or major protocol deviations.
Measure: Median (95% Confidence Interval); unit: log₂ titer
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
log₂ titer
  Day 0 | 56.89 [36.00 to 181.0] | 36.00 [22.63 to 90.51]
  Day 28 | 1152.1 [576.0 to 1448.2] | 724.1 [362.0 to 1152.1]

10. Secondary Outcome: Seroprotection Rate
Description: Seroprotection rate was defined as the percentage of participants in each group with anti-type 2-specific poliovirus neutralizing antibodies titers ≥ 1:8.
Time Frame: Day 0 and Day 28
Population: All randomized participants who received study vaccine and had no exclusion criterion or major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 15
percentage of participants
  Day 0 (pre-vaccination) | 100 [78.2 to 100] | 93.3 [68.1 to 99.8]
  Day 28 | 100 [78.2 to 100] | 100 [78.2 to 100]

11. Secondary Outcome: Seroconversion Rate
Description: Seroconversion rate is defined as the percentage of participants in each group with a change from seronegative to seropositive (poliovirus type-2-specific neutralizing antibody titers ≥ 1:8) or, in participants seropositive at Baseline, an increase in neutralizing antibody titer of at least four-fold from Baseline.
Time Frame: Day 28
Population: Randomized participants who received study vaccine with no exclusion criterion or major protocol deviations. Five participants (2 in the nOPV2-Candidate 1 group, 3 in the nOPV2-Candidate 2 group) with pre-vaccination type 2- neutralizing antibody titers too close to the upper limit of quantitation to measure a 4-fold increase are excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 12 | 13
percentage of participants | 83.3 [51.6 to 97.9] | 84.6 [54.6 to 98.1]

12. Secondary Outcome: Neurovirulence Assessed by the Average Percent Paralysis in Inoculated Mice
Description: Neurovirulence of shed virus was measured using a modified WHO poliovirus receptor transgenic mouse neurovirulence test (mTgmNVT). The last stool sample provided by each participant that had adequate concentrations of virus for the neurovirulence assay (≥ 4 log₁₀[CCID₅₀/g]) was used in the test. For each stool specimen thirty Tg-PVR21 mice were administered intraspinal inoculations of 4 log₁₀(CCID₅₀) amplified virus. After 14 days the inoculated mice were assessed as either paralyzed or non-paralyzed. For each participant/sample, the percentage of paralyzed mice was calculated. Overall percent paralysis is the average percentage of paralyzed mice over all participants in each group.
Time Frame: Samples tested were the last post-vaccination sample per participant suitable for analysis; samples used in the analysis ranged from Day 2 to Day 56
Population: Participants with stool samples evaluable by the neurovirulence test; in the nOPV2-Candidate 2 group only six participants shed sufficient virus at any time point to attempt virus amplification, and amplification did not work for four of these.
Measure: Mean (Full Range); unit: percent paralysis
Units Other Than Participants: innoculated mice
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
Number analyzed (Participants) | 15 | 2
Number analyzed (innoculated mice) | 446 | 58
percent paralysis | 1.6 [0.0 to 10] | 6.9 [0.0 to 14.3]

ADVERSE EVENTS:
Time Frame: From Day 0 up to 42 days
Arm/Group | Novel OPV2 Candidate 1 | Novel OPV2 Candidate 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Novel OPV2 Candidate 1 (N=15) | Novel OPV2 Candidate 2 (N=15)
Blood creatine phosphokinase increased (Investigations) | 9 | 11
Aspartate aminotransferase increased (Investigations) | 7 | 9
Alanine aminotransferase increased (Investigations) | 6 | 8
Bilirubin conjugated increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 5
Syncope (Nervous system disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Enterobiasis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Root canal infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Nervousness (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03430349/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03430349/SAP_001.pdf